CLINICAL TRIAL: NCT01952379
Title: Inflammation in Melasma: Study of Its Infiltrate and the Expression of Acute and Chronic Mediators
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Dermatology department research director, Universidad Autonoma de San Luis Potosí
Other Study IDs: mel-Infla1
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Melasma
Keywords: Melasma; Lymphocytes; Macrophages; Mast cells; Interleukin 17; COX-2; Inflammation
MeSH Terms: conditions — Melanosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 3 mm Skin punch biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Melasma: Women affected by symmetric facial malar melasma.

SUMMARY:
Melasma is an acquired hyperpigmentary disorder that commonly affects women from Asia and Latin-America.There is evidence of subclinical inflammation supported by diffuse spectrometry and by prominent inflammatory cells in affected areas; however this infiltrate and its inflammatory mediators remains unexplored. Chronic inflammation induces melanogenesis and angiogenesis; thus, it could be linked to its recurrent nature.Therefore, the aim of this study is to describe the inflammatory cellular infiltrate, and the expression of main inflammatory and angiogenic mediators in this condition, as well as to explore its relationship with severity of disease.

Using histological, histochemistry, immunohistochemistry, and quantitative real-time PCR, we evaluated melasma lesions from 20 healthy female patients with malar melasma without specific solar exposure or photoprotection measures within the previous 3 weeks and compared them to non lesional skin.

DETAILED DESCRIPTION:
Melasma is a frequent, photoinduced, pigmentary disorder among latin-american women. Its etiology is not completely elucidated; however, there is evidence of a melanogenic paracrine cytokine network between the melanocyte and other skin cells, including keratinocytes, fibroblasts, vascular and inflammatory cells, which regulate melanocyte function.

Previous reports in lesional skin have described increased mast cell infiltration in elastotic areas, presence of a moderate lymphohistiocytic infiltrate, increased vascularity, and up-regulation of proangiogenic factors. This histological evidence of skin inflammation is also supported clinically by colorimetry and thermography, and by the improvement of pigmentation with topical anti-inflammatories.

Photoinduced dermal inflammation might be related to epidermal hyperpigmentation through the production of melanogenic cytokines, and growth factors, and through the secretion of COX-2 induced prostaglandins by keratinocytes, a mechanism involved in the pathogenesis of postinflammatory hyperpigmentation which has not been evaluated in melasma.

The aim of this study is to describe the ongoing characteristics of inflammation in this condition by measuring the cellular infiltrate, the expression of acute and chronic immune inflammatory mediators, and non-immune inflammation mechanism such as COX-2, as well as to explore its relationship with severity of disease, elastosis, and melanin staining.

Twenty healthy female patients with malar melasma without specific solar exposure or photoprotection measures within the previous 3 weeks were enrolled. Disease severity was estimated using the Melasma Area and Severity Index (MASI). Histological, histochemical, immunohistochemistry, and quantitative real-time PCR were used to evaluate the presence of these markers in melasma lesions and compare them to nonlesional skin.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years under signed informed consent form.
* Symmetrical and bilateral lesions.
* Melasma with MASI scores greater than 12 points.

Exclusion Criteria:

* Melasma treatment or photoprotection measures within last 2 months.
* Pregnant women or nursing.
* Miscarriage or labor in the last 12 months.
* Menopause
* Coexistence of other pigmentation disorders.
* Infrared radiation exposure.
* Regular exercise or diet restriction.
* Consumption of food supplements.
* Any type of drugs consumption in the last 2 months (i.e anti-inflammatories and hormonal treatments)
* Personal history of keloid or hypertrophic scars.
* Lidocaine allergy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women affected with malar melasma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Inflammatory cellular infiltrate | Single time measurement
  Determine by immunohistochemistry common inflammatory cellular infiltrate in melasma lesions and non affected skin (i.e CD1, CD68, CD4, CD8).

SECONDARY OUTCOMES:
Acute inflammatory mediators | Single time measurement
  Determine by immunohistochemistry, and PCR techniques, the expression of IL1 alpha, IL1 beta, IL1 alpha receptor, and VEGF in melasma lesions and non affected skin.
Chronic inflammatory mediators | Single time measurement
  Determine by immunohistochemistry, and PCR techniques, the expression of COX-2, and IL-17 in melasma lesions and non affected skin.

OTHER OUTCOMES:
Correlation between inflammation markers and pigmentation | Single time measurement
  Analyze inflammation parameters and to correlate data with melanin, elastosis, and clinical parameters of severity.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castanedo-Cazares, MD, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"; Bertha Torres-Alvarez, MD, Study Chair — Hospital Central "Dr. Ignacio Morones Prieto"; Adriana Rodriguez-Arambula, MD, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Navarrete-Solis J, Castanedo-Cazares JP, Torres-Alvarez B, Oros-Ovalle C, Fuentes-Ahumada C, Gonzalez FJ, Martinez-Ramirez JD, Moncada B. A Double-Blind, Randomized Clinical Trial of Niacinamide 4% versus Hydroquinone 4% in the Treatment of Melasma. Dermatol Res Pract. 2011;2011:379173. doi: 10.1155/2011/379173. Epub 2011 Jul 21. PMID 21822427
- [Background] Torres-Alvarez B, Mesa-Garza IG, Castanedo-Cazares JP, Fuentes-Ahumada C, Oros-Ovalle C, Navarrete-Solis J, Moncada B. Histochemical and immunohistochemical study in melasma: evidence of damage in the basal membrane. Am J Dermatopathol. 2011 May;33(3):291-5. doi: 10.1097/DAD.0b013e3181ef2d45. PMID 21317614
- [Background] Moncada B, Sahagun-Sanchez LK, Torres-Alvarez B, Castanedo-Cazares JP, Martinez-Ramirez JD, Gonzalez FJ. Molecular structure and concentration of melanin in the stratum corneum of patients with melasma. Photodermatol Photoimmunol Photomed. 2009 Jun;25(3):159-60. doi: 10.1111/j.1600-0781.2009.00425.x. PMID 19438997
- [Background] Hernandez-Barrera R, Torres-Alvarez B, Castanedo-Cazares JP, Oros-Ovalle C, Moncada B. Solar elastosis and presence of mast cells as key features in the pathogenesis of melasma. Clin Exp Dermatol. 2008 May;33(3):305-8. doi: 10.1111/j.1365-2230.2008.02724.x. PMID 18419607
- [Background] Espinal-Perez LE, Moncada B, Castanedo-Cazares JP. A double-blind randomized trial of 5% ascorbic acid vs. 4% hydroquinone in melasma. Int J Dermatol. 2004 Aug;43(8):604-7. doi: 10.1111/j.1365-4632.2004.02134.x. PMID 15304189